CLINICAL TRIAL: NCT06649396
Title: Determination of New Detection and Quantification Thresholds for Serological and Molecular Tests for Hepatitis Delta Virus (HDV) Using Capillary Blood on Blotting Paper (DBS)
Acronym: SACADE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: CNR Hepatite Delta (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMEA
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Delta Hepatitis
Keywords: Dried Blood Spot; DBS; Delta Hepatitis; HDV; Viral load; Serology
MeSH Terms: conditions — Hepatitis D | interventions — Dried Blood Spot Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capillary Blood on DBS (Experimental): A total of 100µL of capillary blood will be deposited onto DBS
  Interventions: Diagnostic Test: Dried Blood Spot
- Plasma from EDTA whole blood (Experimental): Plasma from peripheral blood
  Interventions: Diagnostic Test: Analysis on plasma

INTERVENTIONS:
Diagnostic Test: Dried Blood Spot — Comparing analysis results between dried blood spot and plasma
  Arms: Capillary Blood on DBS
Diagnostic Test: Analysis on plasma — Analysis on plasma
  Arms: Plasma from EDTA whole blood

SUMMARY:
The Delta hepatitis virus (HDV) is a satellite virus that requires the presence of hepatitis B virus (HBV) for infection. Approximately 5% of HBV-infected individuals, or about 12 million people globally, are also carriers of HDV. This dual infection significantly heightens the risk of liver damage and the progression to hepatocellular carcinoma (HCC).

Historically, the diagnosis of HDV has been limited, leading to an underestimation of its true prevalence both nationally and internationally. Recent advancements in treatments for viral hepatitis and the introduction of new HDV-specific therapies have spurred increased interest in the virus, prompting public health authorities to call for improved diagnostic and monitoring tools.

Detection of HDV typically involves serological tests (ELISA/CLIA) on serum or plasma, followed by viral load quantification using RT-qPCR if positive. However, laboratory access is often insufficient in many regions, particularly affecting marginalized populations and high-endemic areas, especially in low-resource countries. New sample collection methods that help connect patients to expert laboratories are needed, as shipping frozen biological samples can be complex and costly.

In response, Dried Blood Spot (DBS) sampling-where serum, plasma, or whole blood is dried on filter paper-has been adopted by numerous public health organizations as a simple, cost-effective, and non-infectious means of storage and transport. DBS is already validated for diagnosing and monitoring infections such as HIV, HBV, and HCV.

Given the unique biology of each virus, specific studies are required to determine how using DBS affects detection and quantification thresholds for each laboratory technique. The National Reference Center for Delta Hepatitis (CNR-Delta), commissioned by Public Health France, has developed a DBS protocol for HDV, based on available literature and prior studies regarding storage conditions and reconstitution solutions. Two retrospective studies utilizing CNR collections have established new positivity thresholds for serology and detection/quantification in molecular biology for serum/plasma and EDTA whole blood on DBS.

To finalize this protocol, further study of thresholds for capillary blood tests on DBS is essential. Capillary blood, obtained via finger prick, could simplify the use of this tool, reducing the need for specialised equipment and expertise, and potentially allowing for self-sampling by patients.

The current study aims to validate the DBS tool for HDV serological and molecular testing using capillary blood. The hypothesis posits that geographical barriers to accessing hospitals and laboratories for HDV patients complicate the shipping of frozen plasma samples, increasing costs. Developing a serological screening and viral load testing technique from a drop of capillary blood on DBS paper could effectively link patients to specialized centers. Since DBS is considered non-infectious, it also mitigates administrative complications.

By comparing results from paired samples-plasma (the gold standard) from EDTA whole blood and capillary blood on DBS-we aim to redefine detection and quantification thresholds for both methods. Validating these new thresholds will allow the use of this tool while maintaining quality standards for diagnosing and monitoring active HDV infections.

DETAILED DESCRIPTION:
The Delta hepatitis virus (HDV) is a satellite virus that requires the presence of hepatitis B virus (HBV) for infection. Approximately 5% of HBV-infected individuals, or about 12 million people globally, are also carriers of HDV. This dual infection significantly heightens the risk of liver damage and the progression to hepatocellular carcinoma (HCC).

Historically, the diagnosis of HDV has been limited, leading to an underestimation of its true prevalence both nationally and internationally. Recent advancements in treatments for viral hepatitis and the introduction of new HDV-specific therapies have spurred increased interest in the virus, prompting public health authorities to call for improved diagnostic and monitoring tools.

Detection of HDV typically involves serological tests (ELISA/CLIA) on serum or plasma, followed by viral load quantification using RT-qPCR if positive. However, laboratory access is often insufficient in many regions, particularly affecting marginalized populations and high-endemic areas, especially in low-resource countries. New sample collection methods that help connect patients to expert laboratories are needed, as shipping frozen biological samples can be complex and costly.

In response, Dried Blood Spot (DBS) sampling-where serum, plasma, or whole blood is dried on filter paper-has been adopted by numerous public health organizations as a simple, cost-effective, and non-infectious means of storage and transport. DBS is already validated for diagnosing and monitoring infections such as HIV, HBV, and HCV.

Given the unique biology of each virus, specific studies are required to determine how using DBS affects detection and quantification thresholds for each laboratory technique. The National Reference Center for Delta Hepatitis (CNR-Delta), commissioned by Public Health France, has developed a DBS protocol for HDV, based on available literature and prior studies regarding storage conditions and reconstitution solutions. Two retrospective studies utilizing CNR collections have established new positivity thresholds for serology and detection/quantification in molecular biology for serum/plasma and EDTA whole blood on DBS.

To finalize this protocol, further study of thresholds for capillary blood tests on DBS is essential. Capillary blood, obtained via finger prick, could simplify the use of this tool, reducing the need for specialised equipment and expertise, and potentially allowing for self-sampling by patients.

The current study aims to validate the DBS tool for HDV serological and molecular testing using capillary blood. The hypothesis posits that geographical barriers to accessing hospitals and laboratories for HDV patients complicate the shipping of frozen plasma samples, increasing costs. Developing a serological screening and viral load testing technique from a drop of capillary blood on DBS paper could effectively link patients to specialized centers. Since DBS is considered non-infectious, it also mitigates administrative complications.

By comparing results from paired samples-plasma (the gold standard) from EDTA whole blood and capillary blood on DBS-we aim to redefine detection and quantification thresholds for both methods. Validating these new thresholds will allow the use of this tool while maintaining quality standards for diagnosing and monitoring active HDV infections.

The benefits of the capillary blood on DBS protocol include:

* For patients: Improved access to care regardless of geographic location and easier sampling (self-sampling).
* For clinicians: Simplified management and extended screening to hard-to-reach populations.
* For laboratories: Reduced transportation costs and infectious risk.
* For the CNR: The opportunity to study global prevalence with a simplified protocol.

In summary, the "gold standard" for diagnosing and monitoring HDV infection involves serology on serum or plasma, testing for total anti-HDV antibodies followed by viral load quantification. To assess whether tests from dried capillary blood can replace plasma/serum tests, a comparative study is necessary, where plasma samples and a drop of capillary blood are collected simultaneously from the same patient and tested in parallel. This comparison will evaluate the sensitivity and specificity of the DBS tool using capillary blood and establish new detection and quantification thresholds for viral load on DBS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years old and above)
* Patient infected by the Hepatitis Delta Virus (HDV positive serology)
* Patient followed by one of the participating APHP hospitals' hepatology department
* Patient for whom peripheral blood sampling is already planned as part of their medical follow-up.
* Free, informed and signed consent.

Exclusion Criteria:

* Patient without blood sampling scheduled as part of medical follow-up.
* Patient with a condition that makes fingertip capillary puncture impossible.
* Patient refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
HDV serology | At enrollment
  Comparison between total anti-HDV antibody detection results on Diasorin Liaison XL on plasma obtained from peripheral blood (EDTA) and on capillary blood blotted onto filter paper.
HDV viral load | At enrollment
  Comparison between HDV viral load results obtained by RT-qPCR (Eurobioplex EBX-071) on plasma from peripheral blood (EDTA) and capillary blotted onto filter paper.

SECONDARY OUTCOMES:
Genotyping | At enrollment
  Comparison between R0 RNA sequences (SANGER) on plasma obtained from peripheral blood (EDTA) and capillary blood blotted onto filter paper.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre National de Référence associé de l'Hépatite Delta (CNR-Delta), Bobigny, France

IPD SHARING:
Plan to Share IPD: No
All data will anonymous